CLINICAL TRIAL: NCT00424749
Title: A Pilot Study on the Use of Rituximab in the Treatment of Churg- Strauss Syndrome With Renal Involvement
Brief Title: Rituxan in Churg Strauss Syndrome With Renal Involvement
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company providing study drug terminated study due to lack of funds
Sponsor: Fernando Fervenza (Other)
Collaborators: Genentech, Inc. (Industry); Biogen (Industry); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Fernando Fervenza, MD, PhD, Professor of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-004767; UL1RR024150 (NIH)
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-11

CONDITIONS: Churg-Strauss Syndrome
Keywords: Antineutrophil cytoplasmic antibody associated vasculitis; Glomerulonephritis; Rituximab
MeSH Terms: conditions — Churg-Strauss Syndrome; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Glomerulonephritis | interventions — Rituximab; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab (Experimental): 375 mg/m^2/week for 4 weeks
  Interventions: Drug: Rituximab; Drug: Prednisone

INTERVENTIONS:
Drug: Rituximab — Patients received 4 weekly doses of rituximab 375 mg/m^2.
  Other Names: Rituxan; MabThera
Drug: Prednisone — Prednisone 1 mg/kg/day (not to exceed 80 mg/day) for 4 weeks followed by a taper to 0 mg by 6 months
  Other Names: Deltasone; Liquid Pred; Meticorten; Orasone; Prednicen-M; Prednicot; Sterapred; Sterapred DS

SUMMARY:
Churg-Strauss Syndrome (CSS) is a disease characterized by asthma, abnormally high amounts of eosinophils (a type of white blood cell), and blood vessel inflammation. About 25% of CSS patients develop kidney disease. The goal of this pilot study was to evaluate the safety and effectiveness of Rituximab in inducing remission of kidney disease in patients with CSS.

DETAILED DESCRIPTION:
Churg-Strauss syndrome (CSS) is a small vessel systemic vasculitis associated with asthma and eosinophilia that causes glomerulonephritis in about 25% of patients. Rituximab is a chimeric anti-CD20 monoclonal antibody that depletes B cells and is effective in numerous autoimmune disease including antineutrophil cytoplasmic antibody (ANCA)-associated vasculitis. The aim of this study was to evaluate the safety and efficacy of Rituximab in inducing remission of renal disease activity in patients with CSS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Churg-Strauss syndrome as defined by meeting one of 3 sets of criteria for Churg-Strauss Syndrome described above who have not yet been treated, who have failed steroid therapy (partial or non-responders) or who can not been tapered off oral prednisone because of documented relapsing disease
* Renal involvement (>25% dysmorphic red cell, red blood cell casts, or pauci-immune glomerulonephritis on biopsy)
* Age >18 years old
* Serum creatinine less than or equal to 3.0 mg/dl
* Able and willing to give written informed consent and comply with the requirements of the study protocol.
* Negative serum pregnancy test (for women of child bearing age)
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months after completion of treatment.

Exclusion Criteria

* Severe obstructive or restrictive lung disease (forced expiratory volume in one second <1)
* Cerebral involvement
* Rapidly progressive optic neuropathy or retinal vasculitis
* Active gastrointestinal bleeding
* Heart failure, including pericarditis or myocarditis.
* Hemoglobin <8.5 gm/dL
* Platelets <100,000/mm
* AST or ALT >2.5 Upper Limit of Normal unless related to primary disease
* Positive Hepatitis B or C serology
* History of positive HIV testing
* Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
* Previous treatment with Rituximab
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History of recurrent significant infection or history of recurrent bacterial infections
* Known active bacterial, viral fungal mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* Lack of peripheral venous access
* History of drug, alcohol, or chemical abuse within 6 months prior to screening
* Pregnancy or lactation
* Concomitant malignancies or previous malignancies, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease)
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando C. Fervenza, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Cartin-Ceba R, Keogh KA, Specks U, Sethi S, Fervenza FC. Rituximab for the treatment of Churg-Strauss syndrome with renal involvement. Nephrol Dial Transplant. 2011 Sep;26(9):2865-71. doi: 10.1093/ndt/gfq852. Epub 2011 Feb 16. PMID 21325353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was done between June 2007 and July 2009. Participants were enrolled at the Mayo Clinic in Rochester, MN.
Period: Overall Study
Arm/Group | Rituximab
Started | 4
Completed | 3
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Secondary Outcome: Participants With Normalization of Eosinophil Count at 6 Months
Description: Normalization of eosinophil counts was defined as total eosinophil counts <1.5 x 10^9/L.
Time Frame: 6 months after beginning of remission induction regimen
Measure: Number; unit: participants
Groups:
- Rituximab: The remission induction regimen included oral prednisone and rituximab. Prednisone was started at 1 mg/kg/day for 4 weeks followed by a taper to 0 mg by 6 months. Rituximab 375 mg/m2 intravenously, once a week for 4 weeks was given within 2 weeks of starting steroid therapy.
Arm/Group | Rituximab
Number analyzed (Participants) | 3
participants | 2

2. Primary Outcome: Participants With Remission of Renal Disease Activity at 3 Months
Description: Remission of renal disease activity was indicated by stable or falling creatinine, absence of active urinary sediment AND reduction of oral prednisone dose to less than 50% of average dose of preceding 3 months or less than 10 mg/day (whichever smaller)
Time Frame: 3 months after beginning of remission induction regimen
Measure: Number; unit: participants
Arm/Group | Rituximab
Number analyzed (Participants) | 3
participants | 3

ADVERSE EVENTS:
Time Frame: 1 year after beginning of the remission induction regimen
Description: Safety was assessed by monitoring and recording of adverse events, defined as any untoward medical occurrences in a patient participating in the trial, regardless of causality assessment.
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=3)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Participant was treated with oral antibiotic therapy and recovered.

LIMITATIONS AND CAVEATS:
The limited number of individuals enrolled into the study makes it difficult to draw firm conclusions that are more than hypothesis generating. The company providing study drug terminated study due to lack of funds.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No